CLINICAL TRIAL: NCT04069351
Title: Body Composition Changes During Overfeeding Plus Resistance Training: Influence of Rate of Mass Gain, Assessment Method, and Participant Standardization
Brief Title: Body Composition Changes During Overfeeding Plus Resistance Training
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Texas Tech University (Other)
Collaborators: Dymatize Enterprises, LLC (Unknown); MuscleSound (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: IRB2019-356
Record Dates: First submitted 2019-08-14; First posted 2019-08-28 (Actual); Last update posted 2020-05-07 (Actual); Status verified 2020-05

CONDITIONS: Weight Gain; Resistance Training; Overeating
MeSH Terms: conditions — Weight Gain; Hyperphagia | interventions — Resistance Training

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Overfeeding Plus Resistance Training Arm (Experimental): 6-week overfeeding plus resistance training arm
  Interventions: Dietary Supplement: High-calorie mass gainer supplement; Other: Resistance Training

INTERVENTIONS:
Dietary Supplement: High-calorie mass gainer supplement — A high-calorie mass gainer supplement will be provided to all participants to promote weight gain.
Other: Resistance Training — All participants will complete a 6-week supervised resistance training program.

SUMMARY:
This study will examine the relationship between the rate and composition of mass gain during overfeeding plus resistance training, investigate the validity of multiple assessment methods for quantifying body composition changes during this period, and evaluate the effects of subject presentation on the interpretation of body composition changes.

DETAILED DESCRIPTION:
This study will examine the relationship between the rate and composition of mass gain during overfeeding plus resistance training, investigate the validity of multiple assessment methods for quantifying body composition changes during this period, and evaluate the effects of subject presentation on the interpretation of body composition changes. For this study, resistance-trained males between the ages of 18 and 40 will be recruited. At baseline, participants will complete body composition and metabolism assessments after an overnight period of fasting and resting (i.e. standardized conditions). These baseline assessments will be repeated in the afternoon of the same day after a period of ad libitum physical activity and dietary intake (i.e. non-standardized conditions). At both visits, body composition will be evaluated by a criterion 4-compartment model, necessitating assessments via dual-energy x-ray absorptiometry, air displacement plethysmography, and bioimpedance spectroscopy. Additional assessments will be conducted using single- and multi-frequency bioelectrical impedance analysis, infrared 3-dimensional scanning, and ultrasonography. At a separate baseline session, muscular performance will be measured via 1-repetition maximum and repetitions-to-failure tests on the barbell bench press and plate-loaded hip sled. Once baseline assessments are completed, participants will commence a 6-week, 3-days/week, full-body, progressive resistance training intervention in conjunction with overfeeding. During the intervention, participants will be asked to maintain their habitual diet while also consuming a high-calorie protein/carbohydrate supplement designed to promote mass gain. Dietary recommendations to promote adequate protein intake for maximal fat-free mass accretion will also be provided. For all participants, a target mass gain of 1+ pounds per week will be implemented. However, due to known variability in the propensity to gain body mass during overfeeding and resistance training, it is expected that natural variability in the actual mass gained will be present at the conclusion of the study. After the overfeeding plus resistance training intervention is completed, participants will complete three post-intervention research visits, which will be identical to the baseline visits. Appropriate statistical methods will be used to address the specific aims of this project. These will include linear regression analysis, paired-samples t-tests, effect size calculations, and validity evaluation through metrics such as the constant error, total error, standard error of the estimate, and 95% limits of agreement.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 18 and 40
* Male
* Generally healthy (defined as an absence of any disease or medical condition which could potentially be impacted by study participation, including but not limited to cardiac, musculoskeletal, pulmonary, renal, immunological, or metabolic diseases)
* Weight-stable (defined as no change in body mass >5 pounds [2.3 kg] in the past 3 months)
* Willingness to adhere to study protocol, particularly the completion of the supervised resistance training program and consumption of dietary supplements
* Desire and/or willingness to attempt to gain body mass as part of study intervention
* Resistance trained (defined as performance of resistance training on 2 to 5 days for at least 6 months prior to study initiation), as well as meeting the objective criteria below
* Maximal strength > 1.0 x body mass on the barbell bench press exercise, executed with proper form
* Maximal strength > 2.0 x body mass on plate-loaded hip sled, executed with proper form

Exclusion Criteria:

* Failing to meet any of the aforementioned inclusion criteria
* Height greater than 75.5 inches (due to height limitation of DXA scanner)
* Weight greater than 350 pounds (due to weight limitation of DXA scanner)
* Beard longer than ½ inch (and unwillingness to shave) due to the impact of facial hair on Bod Pod body volume estimates
* History of anabolic-androgenic steroid use, based on self-report

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2019-09-18 (Actual); Primary Completion 2019-11-26 (Actual); Study Completion 2019-11-26 (Actual)

PRIMARY OUTCOMES:
Proportion of Body Mass Gained as Fat-Free Mass | 6 weeks
  Calculated as change in fat-free mass (in kilograms) divided by change in body mass (in kilograms).
Rate of Body Mass Gain | 6 weeks
  Rate of body mass gained calculated in kilograms gained per week.
Fat-free mass | 6 weeks
  Fat-free mass in kilograms, assessed via multiple methods.
Fat mass | 6 weeks
  Fat mass in kilograms, assessed via multiple methods.
Skeletal muscle size | 6 weeks
  Muscle thickness in centimeters.
Resting metabolism | 6 weeks
  Resting metabolism in kcal/day.
Body mass | 6 weeks
  Body mass in kilograms

SECONDARY OUTCOMES:
Muscular Strength (1-repetition maximum test) | 6 weeks
  Maximal muscular strength in kilograms as assessed by 1-repetition maximum test.
Muscular Endurance (repetitions until failure) | 6 weeks
  Muscular endurance in repetitions (i.e. repetitions until failure) using a sub-maximal load.
Skeletal Muscle Quality via Ultrasonography | 6 weeks
  Skeletal muscle quality via ultrasonography (e.g. echo intensity in arbitrary units).
Estimated Skeletal Muscle Glycogen | 6 weeks
  Estimated muscle glycogen as assessed via ultrasound, in arbitrary units.
Estimated Skeletal Muscle Intramuscular Fat | 6 weeks
  Estimated intramuscular fat as assessed via ultrasound, in arbitrary units

CONTACTS AND LOCATIONS:
Locations (1):
- Texas Tech University, Lubbock, Texas, United States

REFERENCES:
- [Derived] Rodriguez C, Harty PS, Stratton MT, Siedler MR, Smith RW, Johnson BA, Dellinger JR, Williams AD, White SJ, Benavides ML, Tinsley GM. Comparison of Indirect Calorimetry and Common Prediction Equations for Evaluating Changes in Resting Metabolic Rate Induced by Resistance Training and a Hypercaloric Diet. J Strength Cond Res. 2022 Nov 1;36(11):3093-3104. doi: 10.1519/JSC.0000000000004077. Epub 2021 Jun 22. PMID 34172636